CLINICAL TRIAL: NCT00400907
Title: Follow-up Observational Study of the Randomised Intergroup Trial of First Line Treatment for Patients With Diffuse Large B-Cell Non-Hodgkin's Lymphoma With CHOP-Like Chemotherapy Regimen With or Without the Anti-CD20 Antibody Rituximab (IDEC-C2B8) [MINT]
Brief Title: Observation in Patients With Diffuse Large B-Cell Non-Hodgkin's Lymphoma Treated on Clinical Trial CAN-NCIC-LY9
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: German High-Grade Non-Hodgkin's Lymphoma Study Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000514350; DSHNHL-MINT-FU; EU-20656; DSHNHL-M39045
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2007-01

CONDITIONS: Long-term Effects Secondary to Cancer Therapy in Adults; Lymphoma
Keywords: long-term effects secondary to cancer therapy in adults; stage I adult diffuse large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Watchful Waiting

INTERVENTIONS:
Other: clinical observation
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Treatment for diffuse large B-cell non-Hodgkin's lymphoma may cause side effects and secondary cancers later in life. An observational study that evaluates patients after undergoing six courses of combination chemotherapy with or without rituximab and radiation therapy may help doctors predict a patient's response to this treatment and help plan the best treatment.

PURPOSE: This observational study is evaluating patients with diffuse large B-cell non-Hodgkin's lymphoma to see how well treatment on clinical trial CAN-NCIC-LY9 works.

DETAILED DESCRIPTION:
OBJECTIVES:

* Gain information on the long-term efficacy of 6 courses of CHOP (cyclophosphamide, doxorubicin hydrochloride, prednisone, and vincristine)-like chemotherapy with vs without rituximab (plus involved-field radiotherapy to primary bulky disease) in young patients with good-prognosis diffuse large B-cell non-Hodgkin's lymphoma treated on protocol CAN-NCIC-LY9.
* Gain information on late toxicities, including secondary neoplasm occurring in young good-prognosis patients treated on protocol CAN-NCIC-LY9.

OUTLINE: This is a multicenter study.

Patients successfully completing treatment on protocol CAN-NCIC-LY9 are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 667 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients recruited for protocol CAN-NCIC-LY9 and evaluated in the first planned final analysis as of June 2005

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 667 (Estimated)
Dates: Start 2006-01

PRIMARY OUTCOMES:
Time to treatment failure

SECONDARY OUTCOMES:
Complete remission rate
Relapse rate
Overall survival
Tumor control
Disease-free survival
Time to progression
Time to relapse
Late toxicities, particularly organ function deficiencies (e.g., cardiomyopathies), infections, and secondary neoplasms

CONTACTS AND LOCATIONS:
Overall Officials: Michael G.M. Pfreundschuh, MD, Study Chair — Universitaetsklinikum des Saarlandes

REFERENCES:
- [Result] Pfreundschuh M, Kuhnt E, Trumper L, Osterborg A, Trneny M, Shepherd L, Gill DS, Walewski J, Pettengell R, Jaeger U, Zinzani PL, Shpilberg O, Kvaloy S, de Nully Brown P, Stahel R, Milpied N, Lopez-Guillermo A, Poeschel V, Grass S, Loeffler M, Murawski N; MabThera International Trial (MInT) Group. CHOP-like chemotherapy with or without rituximab in young patients with good-prognosis diffuse large-B-cell lymphoma: 6-year results of an open-label randomised study of the MabThera International Trial (MInT) Group. Lancet Oncol. 2011 Oct;12(11):1013-22. doi: 10.1016/S1470-2045(11)70235-2. Epub 2011 Sep 21. PMID 21940214